CLINICAL TRIAL: NCT03673592
Title: Prospective Non-selection Study to Investigate the Clinical Predictive Value of Chromosome Copy Number Values Consistent With the Presence of Mosaicism Within the Trophectoderm Biopsy (NON-SELECTION MOSAICISM)
Brief Title: Clinical Value of Mosaicism Diagnosis on the Trophectoderm Biopsies
Acronym: NS-MOSAICISM
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Responsible Party: Sponsor
Other Study IDs: IGX14-MOS-AC-18-03
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Aneuploidy; Chromosome Abnormality
Keywords: Mosaicism; PGT-A; Blastocyst biopsy; Aneuploidy testing; Preimplantation genetics
MeSH Terms: conditions — Aneuploidy; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA analysis of each patient's embryos
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Euploid embryos analyzed by PGT-A: Embryos with a normal chromosome copy number. This embryos will be transferred to the uterus.
  Interventions: Diagnostic Test: PGT-A
- Low-grade mosaic embryos (PGT-A): Embryos with a lower aneuploidy percentage (<50%). This embryos will be considered for transfer to the uterus.
  Interventions: Diagnostic Test: PGT-A
- High-grade mosaic embryos (PGT-A): Embryos with a high aneuploidy percentage (50-70%). This embryos will be discarded for transfer.
  Interventions: Diagnostic Test: PGT-A
- Aneuploid embryos analyzed by PGT-A: Embryos with an abnormal number of chromosomes. This embryos will be discarded for transfer.
  Interventions: Diagnostic Test: PGT-A

INTERVENTIONS:
Diagnostic Test: PGT-A — PGT-A will be carried out following the usual clinical practice: Trophectoderm biopsy samples from blastocysts are analyzed by NGS to screen for numerical chromosomal abnormalities.

SUMMARY:
Mosaicism within an embryo is defined as the presence of two or more cell populations with different genotypes. Blastocysts classified as mosaic by Preimplamtation Genetic Testing for Aneuploidy (PGT-A) have been reported to implant less and miscarry more frequently than embryos classified as euploid. Because of the unknown impact of mosaicism on embryo development, these embryos are given low priority and are discarded for transfer. However, recent papers on the transfer of human embryos classified by PGT-A as mosaic suggest that embryos with a low fraction of abnormal cells resulting in viable, chromosomally normal ongoing pregnancies, and high-level mosaics resulting in fewer viable pregnancies, but so far none producing mosaic babies.

The apparent presence of mosaicism in an embryo is used as a selection criteria for embryo transfer (ET), introducing a strong bias in terms of patient prognosis and embryo quality. Additionally, it is also possible that some embryos are incorrectly classified as "mosaic" due to technical variability derived from the processing of a uniform aneuploid embryo.

The aims of this study is to provide evidences about the clinical significance of chromosomal mosaicism in PGT-A cycles by a prospective non-selection based methodology.

DETAILED DESCRIPTION:
One of the most common reasons why in vitro fertilization (IVF) is unsuccessful, or why miscarriages occur, is because of chromosomal abnormalities in the embryo. Embryos with less than 20% aneuploidy are considered as euploid, while those between 20-80% are reported as mosaic, and those over 80% as aneuploid. Embryos with the correct number of chromosomes (euploid) have a higher chance of leading to a successful pregnancy than those with the incorrect number of chromosomes (aneuploid) or mosaics.

Mosaicism within an embryo is defined as the presence of two or more cell populations with different genotypes. Preliminary data suggested that embryos identified as mosaic by Preimplamtation Genetic Testing for Aneuploidy (PGT-A) may have a reduced chance of implantation compared with euploid and may play a significant role in pregnancy loss.

Because of the unknown impact of mosaicism on embryo development, these embryos are given low priority and are discarded for transfer. They are transferred mostly in poor prognosis patients, explaining the reported lower clinical performances. However, other recent data regarding the transfer of embryos diagnosed as mosaic has shown that embryos with a low fraction of abnormal cells may result in viable, chromosomally normal ongoing pregnancies.

The apparent presence of mosaicism in an embryo is used as a selection criteria for embryo transfer (ET), introducing a strong bias in terms of patient prognosis and embryo quality. Additionally, it is also possible that some embryos are incorrectly classified as mosaic due to technical variability derived from the processing of a uniform aneuploid embryo. Thus, there is an urgent need to understand how to appropriately select and counsel patients regarding such embryos.

This study aims to provide evidences about the clinical significance of chromosomal mosaicism in PGT-A cycles by a prospective non-selection based methodology.

The objectives are to investigate the clinical predictive value for intermediate copy number results consistent with the presence of low mosaicism in TE biopsies, and to validate the thresholds for the classification of embryos in relation with their reproductive potential, providing comprehensive data for clinicians and patients. To demonstrate these objectives, a total of 878 participants are expected to be recruited in 18 months. As the datapoints required for comparison concern embryo transfers rather than participants, this number could be lower depending on the number of embryo transfers received by each participant.

ELIGIBILITY:
Inclusion Criteria:

* PGT-A cases for any medical indication and sign the written informed consent form approved by the Ethics Committee (EC) after having been duly informed of the nature of the research and voluntarily accepted to participate in the study.
* Only PGT-A cycles with own oocytes.
* Female age up to 44 years old (also included).
* ICSI treatment must be done in all oocytes.
* Have at least one euploid blastocyst or one low-grade mosaicism diagnosis for a single chromosome after PGT-A analysis (excluding aneuploidies compatible with life, e.g. chromosomes 13, 18, 21 and X/Y).
* Single or Double Embryo Transfer (SET or DET). The patient remains included in the study until the 4th ET (fresh or frozen) from the initial stimulation cycle or until patient's enrolment period ends (whichever comes first). The data collected until one of these points will be included in the study, whilst clinical outcomes from additional ET will be disregarded.

Exclusion Criteria:

* No embryo reaching blastocyst stage with a proper morphology for trophectoderm biopsy.
* Embryo transfer coming from the worst grade blastocyst morphology according to Gardner's criteria (Annex 1) will be excluded.
* DET resulting in singletons. (Note: DET resulting in dizygotic twins or implantation failure to the both embryos transferred will be allowed).
* Any illness or medical condition that is unstable or can put patient safety at risk and compliance in the study.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Embryos from IVF patients up to 44 years of age (also included) undergoing PGT-A.
Study Population: Embryos from In Vitro Fertilization (IVF) patients up to 44 years old (also included) with medical indication of PGT-A and own oocytes.
Sampling Method: Non-Probability Sample
Enrollment: 783 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Sustained implantation rate | 20 weeks after the embryo transfer
  Presence of a viable pregnancy after 20 weeks of gestation measured by ultrasound scan

SECONDARY OUTCOMES:
Miscarriage rate | 20 weeks after the embryo transfer
  The spontaneous loss of an intra-uterine pregnancy prior to 20 completed weeks of gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Capalbo, BSc PhD, Principal Investigator — Igenomix S.L.
Locations (3):
- Italy (3):
  - Demetra, Florence
  - Genera, Roma
  - Humanitas Fertility Center, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capalbo A, Poli M, Rienzi L, Girardi L, Patassini C, Fabiani M, Cimadomo D, Benini F, Farcomeni A, Cuzzi J, Rubio C, Albani E, Sacchi L, Vaiarelli A, Figliuzzi M, Findikli N, Coban O, Boynukalin FK, Vogel I, Hoffmann E, Livi C, Levi-Setti PE, Ubaldi FM, Simon C. Mosaic human preimplantation embryos and their developmental potential in a prospective, non-selection clinical trial. Am J Hum Genet. 2021 Dec 2;108(12):2238-2247. doi: 10.1016/j.ajhg.2021.11.002. Epub 2021 Nov 18. PMID 34798051